CLINICAL TRIAL: NCT05229003
Title: A Randomized, Uncontrolled, Exploratory Phase 2 Trial of Irinotecan Plus Anlotinib or Further in Combination With Penpulimab as Second-line Treatment of Metastatic Colorectal Cancer (ZL-IRIAN)
Brief Title: Irinotecan Plus Anlotinib or Further in Combination With Penpulimab for Second-line Treatment of mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Director of Department of Medical Gastrointestinal Oncology, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-IRIAN
Record Dates: First submitted 2022-01-25; First posted 2022-02-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; second-line treatment; target therapy; enlotinib; penpulimab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — anlotinib; penpulimab; Irinotecan

STUDY DESIGN:
Intervention Model Description: Patients were first enrolled into cohort A, and when the efficacy of cohort A reached a certain percentage, the enrollment of cohort B started then.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cohort A (Experimental): Anlotinib + Irinotecan:
  Anlotinib, 10mg, oral, once daily, D1-10, q2W; Irinotecan, 180mg/m2, iv drip, d6, q2w.
  Interventions: Drug: Anlotinib; Drug: Irinotecan
- cohort B (Experimental): Anlotinib + Penpulimab + Irinotecan:
  Anlotinib, 8mg, oral, once daily, d1-10, q2w; Penpulimab 200mg, i.v. d6, q2w; Irinotecan, 180mg/m2, iv infusion, d6, q2w.
  Interventions: Drug: Anlotinib; Drug: Penpulimab; Drug: Irinotecan

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 8mg or 10mg, d1-9，q2w
Drug: Penpulimab — Penpulimab 200mg, d6, q2w
  Arms: cohort B
Drug: Irinotecan — Irinotecan 180mg/m2, d6, q2w

SUMMARY:
This is an exploratory, non-controlled, multi-cohort, phase II small-sample clinical study designed to evaluate the clinical benefit of second-line treatment with anlotinib plus irinotecan or further in combination with a PD-1 monoclonal antibody (penpulimab) in patients with advanced colorectal cancer after first-line treatment failure. To explore the rationality of the combination of chemotherapy and targeted therapy and immunotherapy strategy and obtain relevant survival and safety data. The study will fully evaluate the efficacy, PFS, OS, safety and related biomarkers of the regimen.

DETAILED DESCRIPTION:
The design of this study is an open, non-controlled, multi-cohort, phase II, small-sample prospective clinical study, including eligible patients with metastatic colorectal cancer who received the second-line treatment, and two cohort were included, Cohort A received anlotinib and irinotecan chemotherapy (n=23), and the treatment of cohort B consisted of anlotinib and anti-PD-1 mab (penpulimab) plus irinotecan chemotherapy. Patients were firstly enrolled in cohort A, and if patients in cohort A achieved an response rate of no less than 15% (i.e., no less than 4 out of 23 patients receiving efficacy evaluation achieved CR/PR), the following patients would be enrolled in cohort B. If the response rate of patients in cohort A was less than 15%, subsequent cohort B enrollment (non-control) would be stopped.

A total of 46 patients enrolled in this study, actually.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent/metastatic colorectal adenocarcinoma confirmed by histopathological pathology report;
2. The patient received oxaliplatin in combination with fluorouracil as the first-line systemic therapy (with or without anti-EGFR mab or VEGF mab) and failed. Fluorouracil (5-FU, capecitabine, or S-1) and oxaliplatin must be included in the first-line regimens. Treatment failure was defined as: disease progression or intolerable toxicity occurred during treatment or within 3 months after the last treatment; Note: Early adjuvant/neoadjuvant therapy is permitted. If recurrence or metastasis occurs during adjuvant/neoadjuvant therapy or within 6 months after completion, adjuvant/neoadjuvant therapy is considered a failure of first-line chemotherapy for advanced disease;
3. With one or more measurable lesions, the longest diameter measured by spiral CT scan should be at least 10 mm, and the longest diameter measured by conventional CT scan should be at least 20 mm (RECIST standard, version 1.1);
4. the type of KRAS, NRAS, BRAF, and MSI were known, requiring wild type of BRAF. Cohort A required patients with MSS/pMMR status.
5. ECOG score was 0-1;
6. Life expectancy ≥12 weeks;
7. The patient has recovered from damage caused by other anti-tumor therapy, received cytotoxic drugs, radiotherapy or surgery for ≥4 weeks, and the wound has completely healed;
8. Bone marrow capacity and liver and kidney function were sufficiently reserved within 7 days before screening: absolute neutrophil (ANC) count ≥1.5x109 /L; Hemoglobin ≥ 8.0g/ dL; Platelet count ≥80 x109 /L; Total bilirubin < 1.5 times upper normal limit (ULN); ALT and AST< 2.5x ULN (with liver metastasis <5x ULN); Serum creatinine ≤1 x ULN, the clearance rate of endogenous creatinine >50ml/min;
9. Women of childbearing age should take effective contraceptive measures;
10. Subjects voluntarily joined the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria:

1. A history of other malignant tumors within 5 years, except cured cervical carcinoma in situ or basal cell carcinoma of the skin;
2. Patients with hypertension that could not be controlled by antihypertensive medication (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg), coronary heart disease of grade I or above, arrhythmia of grade I or above (including prolonged QTc interval > 450ms in males and > 470 ms in females) and cardiac dysfunction of grade I or above;
3. Symptomatic brain or meningeal metastases (unless the patient was treated for >6 months, imaging results were negative within 4 weeks prior to study entry, and tumor-related clinical symptoms were stable at study entry); with a history of uncontrolled epileptic seizures, central nervous system dysfunction, or mental disorders;
4. Uncontrolled pleural or abdominal effusion;
5. Undergoing kidney dialysis;
6. severe or uncontrolled infection;
7. pregnant or lactating women who are fertile but have not taken adequate contraceptive measures;
8. Multiple factors affecting oral medication (inability to swallow, chronic diarrhea and intestinal obstruction);
9. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg< 2G /L), bleeding tendency or receiving thrombolytic or anticoagulant treatment; patients with gastrointestinal bleeding risk should not be enrolled, including the following conditions :(1) active peptic ulcer lesions and fecal occult blood (++); (2) patients with history of black stools and hematemesis within 3 months;
10. Prior exposure to any anti-PD-1 or anti-PD-L1, PD-L2, CD137, CTLA-4 antibody therapy, or any other antibody or drug that specifically targets T-cell costimulation or immune checkpoint pathways.
11. Former treatment of irinotecan for 1 or more cycles;
12. Prior exposure to any anti-VEGFR small molecule inhibitors (e.g. Apatinib, regorafenib, Fruquintinib, Anlotinib, etc.)
13. Participated in clinical trials of other drugs within four weeks
14. Urine routine examination indicated urine protein > 2+, or 24-hour urine protein quantification ≥1.0g/24h
15. Use of immunosuppressive agents within 4 weeks prior to the first dose of study therapy, excluding nasal, inhaled, or other topical or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/ d of prednisone or equivalent doses of other glucocorticoids), or hormone use for the prevention of contrast agent allergy.
16. Residual liver volume is less than 50% of the total liver volume. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | the rate of patients with CR and PR, through study completion, an average of 1 year
  objective response rate

SECONDARY OUTCOMES:
PFS | from the time signing of ICF until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  progression free survival
OS | from the time signing of ICF until the date of death from any cause, assessed up to 36 months
  overall survival
DoR | the time between the first tumor evaluation for CR or PR and the first evaluation for PD(Progressive Disease) or death from any cause, assessed up to 36 months
  duration of response
DCR | the rate of patients with CR, PR and SD, through study completion, an average of 1 year
  disease control rate
AEs | the adverse events rate and types of all enrolled patients, through study completion, an average of 1 year
  the adverse events of all enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China